CLINICAL TRIAL: NCT05179564
Title: Comparison of Different Methods to Assess Glomerular Filtration Rate in Critically Ill Children
Brief Title: Renal Function Assessment in Critically Ill Children
Acronym: IOHEXOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B670201835281
Record Dates: First submitted 2019-03-21; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-10

CONDITIONS: Iohexol; Pharmacokinetics; Renal Function; Critically Ill Children; Acute Kidney Injury; Augmented Renal Clearance
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iohexol plasma clearance (Experimental): a weight-dependent dose of iohexol will be injected as an intravenous bolus in 100 patients
  2,5 -9kg = 1ml; 10-19kg = 2ml; 20-29kg = 3ml; 30-39kg = 4ml; ≥ 40kg = 5ml
  Interventions: Diagnostic Test: iohexol administration; Diagnostic Test: iohexol blood sampling

INTERVENTIONS:
Diagnostic Test: iohexol administration — IV injection of weight-dependent low dose of iohexol at time 0
  Other Names: omnipaque
Diagnostic Test: iohexol blood sampling — Blood sampling will be performed through an arterial (preferred) or venous line, other than the iohexol infusion line. In the first 30 minutes after iohexol injection, a blood sample of 2 ml will be obtained for iohexol concentration measurement and determination of renal biomarkers serum creatinine, cystatin C, betatrace protein. Subsequently, 2 up to 5 additional blood samples of 0,5 ml will be obtained for iohexol determination at 60,120 ,180, 240 and 360 minutes after iohexol injection to calculate iohexol plasma clearance from the plasma disappearance curve

SUMMARY:
Identification of renal dysfunction in critically ill children is often delayed due to lack of accurate methods for evaluation of glomerular filtration rate (GFR). The investigators compared GFR measurement by the gold standard technique iohexol plasma clearance with estimated GFR (eGFR) based on selected established formulas incorporating the renal biomarkers creatinine, cystatin C and betatrace protein.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a frequent comorbidity of critical illness associated with poor outcome, including prolonged duration of mechanical ventilation, longer length of stay and increased mortality or progression to chronic kidney disease on the long term. The reported incidence of AKI in critically ill children and neonates varies widely between 10% and 80% depending on the diagnostic criteria. Besides a decline in renal function, also the phenomenon of augmented renal clearance (ARC) and in consequence enhanced clearance of renally eliminated drugs, is increasingly recognized in pediatric intensive care patients. Hence, accurate assessment of renal function is crucial in the intensive care population to guide therapy. But to date consensus is lacking about the reliability of common GFR estimation methods based on the endogenous renal biomarkers serum creatinine, cystatin C and betatrace protein in critical care patients. the aim of this study is to measure GFR in a reliable way by iohexol plasma clearance and evaluate the agreement between the gold standard technique iohexol plasma clearance and biomarker-based formula to estimate GFR.

ELIGIBILITY:
Inclusion criteria:

* patients admitted to the pediatric or neonatal intensive care unit
* 0 - 15 years
* for neonates: gestational age ≥ 37 weeks
* bodyweight >2.5kg
* intra-arterial and/or intravenous access available for iohexol administration and blood sampling

Exclusion criteria:

* no vascular access in place for iohexol administration and blood sampling
* absence of parental/patient consent
* known hypersensitivity to contrast media or previous history of adverse reaction after administration of contrast agents
* known thyroid dysfunction, or for newborns: mother with known thyroid dysfunction
* extracorporeal circuit (haemodialysis, extra corporal membrane oxygenation (ECMO), peritoneal dialysis)
* patients with chronic kidney disease or congenital kidney anomalies
* preterm neonates (gestational age < 37 weeks)
* body weight < 2.5 kg
* dehydrated newborns (i.e. loss of birth weight ≥ 10%)
* planned/expected surgery with extracorporeal circulation within 5 days after inclusion

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
Agreement between determination of GFR when based on biomarker formulas to estimate GFR compared to measurement of GFR by iohexol plasma clearance | 48 hours
  * GFR will be calculated by using 26 established mathematical equations based on renal biomarkers
  * Iohexol clearance will be calculated from the plasma iohexol disappearance curve based on 3 up to 6 blood samples drawn for iohexol concentration measurement over a 360 minutes interval after iohexol injection, Clearance = iohexol dose /area under the curve
  * Agreement between reference method iohexol clearance and estimating GFR formulas will be evaluated by Bland -Altman analysis with determination of bias (= iohexol clearance - estimated GFR), precision (=standard deviation of bias), limits of agreement (= bias +- 1.96 x standard deviation) and visual display of Bland-Altman plots for every eGFR formula
Identify which GFR estimating formulas yield a sufficient accuracy to predict GFR in critically ill children | 48 hours
  P30 value expresses the percentage of estimated GFR results with evaluated formulas that lie within a 30% range of GFR values measured by iohexol clearance. This P30 value reflects accuracy of a specific GFR estimating formula.
  Formulas with P30 > 75% have acceptable accuracy to be relied on for GFR determination in clinical practice

SECONDARY OUTCOMES:
Prevalence of Acute Kidney Injury and Augmented Renal Clearance based on iohexol clearance in critically ill children | 48 hours
  AKI will be defined by pediatricRIFLE criteria for GFR decline, using age-specific reference values of GFR
  pRIFLE classification of AKI:
  Risk = GFR decline > 25% Injury= GFR decline > 50% Failure= GFR decline > 75%
  ARC will be described as GFR exceeding age-specific reference GFR +2 standard deviations

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Dhont, MD, Principal Investigator — University Hospital, Ghent; Pieter De Cock, PharmD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhont E, Destere A, Gerard A, Bouveyron C, Snauwaert E, Vanhaesebrouck S, De Paepe P, Woillard JB, De Cock P. Accurate Estimation of Glomerular Filtration Rate in Critically Ill Infants and Children Using a Iohexol Population Pharmacokinetic Modeling Approach. Clin Pharmacokinet. 2026 Jan 27. doi: 10.1007/s40262-025-01617-x. Online ahead of print. PMID 41591642
- [Derived] Dhont E, Van Der Heggen T, Snauwaert E, Willems J, Croubels S, Delanghe J, De Waele JJ, Colman R, Vande Walle J, De Paepe P, De Cock PA. Predictors of augmented renal clearance based on iohexol plasma clearance in critically ill children. Pediatr Nephrol. 2024 May;39(5):1607-1616. doi: 10.1007/s00467-023-06221-4. Epub 2023 Nov 23. PMID 37994980
- [Derived] Dhont E, Windels C, Snauwaert E, Van Der Heggen T, de Jaeger A, Dhondt L, Delanghe J, Croubels S, Walle JV, De Paepe P, De Cock PA. Reliability of glomerular filtration rate estimating formulas compared to iohexol plasma clearance in critically ill children. Eur J Pediatr. 2022 Nov;181(11):3851-3866. doi: 10.1007/s00431-022-04570-0. Epub 2022 Sep 2. PMID 36053381